CLINICAL TRIAL: NCT02003846
Title: Comparing the Effects of Bubble Nasal CPAP Versus Ventilator Nasal CPAP in Preterm Infants
Brief Title: Comparing Bubble and Ventilator Nasal CPAP in Preterm Infants
Status: Completed | Type: Observational
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Principal Investigator, Shantanu Rastogi, Attending Neonatologist, Maimonides Medical Center
Other Study IDs: MMC 2013-02-10; MMC 2013-02-10 (Other: Maimonides Medical Center)
Record Dates: First submitted 2013-11-19; First posted 2013-12-06 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Premature infant: Each premature infant will be on bubble nasal CPAP for 2 hours and on ventilator nasal CPAP for 2 hours

SUMMARY:
There are various methods to generate the pressure needed for Nasal CPAP. Some neonatal intensive care units (NICU) use an underwater bubbling system and others use a ventilator to generate the pressure. There is no right or wrong way to generate the pressure and both methods are approved and accepted.

The aim of this study is to compare the two systems of Nasal CPAP by placing the baby on each for a defined time period and reviewing the infant's vital signs. The investigators expect that the pressure generated by bubble CPAP will be better and lead to improved vital signs.

DETAILED DESCRIPTION:
There are various methods to generate the pressure needed for Nasal CPAP. Some neonatal intensive care units (NICU) use an underwater bubbling system and others use a ventilator to generate the pressure. There is no right or wrong way to generate the pressure and both methods are approved and accepted.

The aim of this study is to compare the two systems of Nasal CPAP by placing the baby on each for a defined time period and reviewing the infant's vital signs. The investigators expect that the pressure generated by bubble CPAP will be better and lead to improved vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Neonates between 26-32 weeks gestational age who have been on Nasal CPAP for at least 48hrs on fraction of inspired oxygen (FiO2) of < or = 0.3. Parental consent will be obtained prior to enrollment.

Exclusion Criteria:

* Infants with severe congenital anomalies, such as airway or chest wall deformities, pulmonary hypoplasia, congenital heart disease, neurologic abnormalities including severe intraventricular hemorrhage (IVH) and need for surgery eg. for necrotizing enterocolitis will be excluded from the study. Any infants with genetic/chromosomal abnormalities will be excluded.

Ages: 2 Days to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature infants admitted to the Neonatal Intensive Care Unit (NICU) at Maimonides Medical Center.
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2013-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Physiologic parameters | 2 hours
  heart rate, respiratory rate, oxygen saturation

SECONDARY OUTCOMES:
Physiologic parameters | 2 hours
  cerebral oxygen tissue extraction

CONTACTS AND LOCATIONS:
Overall Officials: Shantanu Rastogi, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

REFERENCES:
- [Background] Gregory GA, Kitterman JA, Phibbs RH, Tooley WH, Hamilton WK. Treatment of the idiopathic respiratory-distress syndrome with continuous positive airway pressure. N Engl J Med. 1971 Jun 17;284(24):1333-40. doi: 10.1056/NEJM197106172842401. No abstract available. PMID 4930602
- [Background] Lee KS, Dunn MS, Fenwick M, Shennan AT. A comparison of underwater bubble continuous positive airway pressure with ventilator-derived continuous positive airway pressure in premature neonates ready for extubation. Biol Neonate. 1998;73(2):69-75. doi: 10.1159/000013962. PMID 9483299